CLINICAL TRIAL: NCT02585050
Title: Influences of DNAR Order Prohibition on Hospital Discharged Ratios and Neurological Outcomes at Discharge
Status: Completed | Type: Observational
Sponsor: Adiyaman University Research Hospital (Other)
Responsible Party: Principal Investigator, Umut Gulacti, Adiyaman University Research Hospital, Adiyaman University Research Hospital
Other Study IDs: ADYU 2
Record Dates: First submitted 2015-10-21; First posted 2015-10-23 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Cardiac Arrest
Keywords: do not attempt resuscitation; neurological outcome; live discharged ratio
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- patients alive discharged from hospital: patients alive discharged from hospital following CPR

SUMMARY:
Debates about the official and legal implementation of Do not attempt resuscitation (DNAR) orders are ongoing. The aim of this study was to determinate factors that influence neurological outcomes at discharge and the ratio of living patients discharged from the hospital due to DNAR prohibition.

DETAILED DESCRIPTION:
Study Design and Setting:

This is a single-center, retrospective chart review performed in a 180-bed rural city hospital.

Methods of Measurements:

Study was conducted as retrospective chart review of CPR call forms that were completed between February 2010 and February 2012. Approximately 450,000 patients were annually admitted to this hospital; 1800 patients were hospitalized in wards, and 500 patients were hospitalized in intensive care units during the study period. A form termed the CPR call form is completed by the leader of the CPR team at the end of all calls. These forms are filed in the hospital archive in chronological order. The hospital uses the resuscitation guidelines from the American Heart Association, and all healthcare providers of the CPR team are certified in basic cardiac life support (BCLS) and advanced cardiovascular life support (ACLS).

Study Population The data were collected from the CPR call forms and hospital medical records. All data were noted by using the Utstein-style reporting template and included the demographic data (date of birth/age and gender), date of arrest, time of first CPR attempt, etiology, preexisting conditions, location of arrest, arrest witnessed (a witnessed cardiac arrest is one that is observed or heard by another person or an arrest that is monitored), initial rhythm, duration of CPR attempt, end of event, date of discharge or death and neurological outcomes at discharge from the hospital.

CPR attempts were defined as an attempt to restore spontaneous circulation by performing chest compressions with or without ventilation. ROSC was defined by a status in which spontaneous circulation was sustained for at least 20 minutes.

Neurological outcomes at discharge were determined with a Cerebral Performance Category (CPC) score based on the last neurological examination of the patients before discharge. CPC scores of 1 or 2 were considered good neurological outcomes, and CPC scores of 3, 4 and 5 were considered poor neurological outcomes.

Data Analysis The continuous variables are expressed as the means and SD. The categorical data are expressed as percentages. Chi-square tests were used for the univariate analyses of categorical variables. Statistical significance was defined as p<0.05. The data were analyzed with SPSS v. 17.0.

ELIGIBILITY:
Inclusion Criteria:

1. Patients experienced inhospital CPR attempts due to cardiac arrest
2. Patients who did not have DNAR orders

Exclusion Criteria:

1. Patients below 18 years of age
2. Calls performed due to code blue drills
3. Missing calls
4. Patients with more than one cardiac arrest
5. Patients with CPR attempts that began outside the hospital who were admitted to the emergency department.
6. Patients with missing the data in hospital medical records.

Ages: 19 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: CPR call forms that were completed.
Sampling Method: Probability Sample
Enrollment: 266 (Actual)
Dates: Start 2010-01; Primary Completion 2012-12 (Actual); Study Completion 2015-01 (Actual)

PRIMARY OUTCOMES:
Examine survival rate from data obtained by retrospective chart review of patients who have not DNAR order and performed CPR due to cardiac arrest in the period 2010-2012 | Two years
  Data obtained by retrospective chart review will data including etiology, preexisting conditions, initial rhythm, end of event (any return of spontaneous circulation or not) live or death at discharged from hospital.

SECONDARY OUTCOMES:
Examine the influence on neurological outcomes at discharge of DNAR order prohibition from data obtained by retrospective chart review. | two years
  Data obtained by retrospective chart review will data including neurological outcomes at discharge from the hospital.

CONTACTS AND LOCATIONS:
Overall Officials: Umut Gulacti, M.D., Principal Investigator — Adiyaman University of Medical Faculty
Locations (1):
- Adiyaman University Research Hospital, Adıyaman, Central, Turkey (Türkiye)

REFERENCES:
- [Result] Field RA, Fritz Z, Baker A, Grove A, Perkins GD. Systematic review of interventions to improve appropriate use and outcomes associated with do-not-attempt-cardiopulmonary-resuscitation decisions. Resuscitation. 2014 Nov;85(11):1418-31. doi: 10.1016/j.resuscitation.2014.08.024. Epub 2014 Sep 4. PMID 25195071